CLINICAL TRIAL: NCT03158012
Title: Evaluation of the Efficacy of an Autologous Microbiome Transplant in Adult Atopic Dermatitis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Richard Gallo, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSD 131244.4
Record Dates: First submitted 2017-05-09; First posted 2017-05-17 (Actual); Results first posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator)
  Interventions: Biological: Autologous Microbial Transplant
- Placebo treatment (Placebo Comparator)
  Interventions: Biological: Autologous Microbial Transplant

INTERVENTIONS:
Biological: Autologous Microbial Transplant — Twice-daily application of Active or Placebo comparators to the right and left ventral arms of patients

SUMMARY:
Unlike healthy control skin, the skin of patients with atopic dermatitis (AD) is frequently colonized by Staphylococcus aureus (S. aureus), putting these patients at increased risk of S. aureus skin infections. In addition, research in the investigator's lab has shown that these patients have fewer protective antimicrobial Staphylococcal species such as Staphylococcal epidermidis (S. epidermidis) that are known to produce antimicrobial peptides that play a role in protecting the skin from invading pathogens. In this study, the investigator will attempt to decrease S. aureus colonization and increase colonization of protective Staph species in AD patients. First the investigator will capture the bacteria on subjects' skin. Next the investigator will selectively grow the subject's antimicrobial Staphylococcal colonies and place them into a base moisturizer. The moisturizer plus bacteria will be applied to one of the subject's arms for one week. Some subjects will receive placebo, which is the moisturizer alone (without bacteria). The investigator will then swab the arms at specified time points during and after the one week application in order to determine whether the S. aureus abundance was affected by the application of the transplanted bacteria.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who are not pregnant or lactating. Female subjects of child-bearing potential must have a negative urine pregnancy test on the day of the screening visit in order to be eligible for the study.
2. 18-60 years of age
3. Diagnosis of atopic dermatitis for at least 6 months using the Hanifin and Rajka Diagnostic Criteria for atopic dermatitis
4. Presence of lesional atopic dermatitis skin in both antecubital fossae
5. Positive S. aureus colonization based on results of a skin culture taken from one of their AD-affected antecubital fossae
6. Positive for antimicrobial CoNS species from non-lesional AD skin

Exclusion Criteria:

1. Use of any topical AD treatments (including topical steroids, topical calcineurin inhibitors) to either arm within one week of the Treatment visit
2. Use of any antihistamines 7 days within one week of the Treatment visit
3. Use of any oral/systemic AD therapies (steroids) within 28 days of the Treatment visit
4. Severe AD that would worsen significantly from holding a participant's usual topical/oral AD medications for the time periods required in the inclusion/exclusion criteria (one week prior to the Treatment visit for topical medications and antihistamines and 28 days prior to Treatment visits for oral medications)
5. Subjects who have taken a bleach bath within a week prior to the Treatment visit, or who take bleach baths during the study
6. Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
7. Subjects with Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier
8. Any subject who is immunocompromised (e.g. provides researchers with a history lymphoma, HIV/AIDS, Wiskott-Aldrich Syndrome) or has a history of malignant disease (with the exception of non-melanomatous skin cancer). This information will be gathered verbally from the patient while taking a medical history from the patient, and will not involve further testing such as an HIV test.
9. Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
10. Active bacterial, viral or fungal skin infections
11. Any noticeable breaks or cracks in the skin on either arm, including severely excoriated skin or skin with open or weeping wounds suggestive of an active infection or increased susceptibility to infection.
12. Ongoing participation in another investigational trial
13. Use of any oral or topical antibiotic for up to four weeks prior to the Treatment visit
14. Use of any systemic immunosuppressive therapy (e.g. CsA, MTX, etc.) within four weeks of the Treatment visit.
15. Sensitivity to or difficulty tolerating Dove fragrance-free bar soap or Cetaphil lotion
16. Subjects with prosthetic heart valves, pacemakers, intravascular catheters, or other foreign or prosthetic devices.
17. Allergy or intolerability to soy or macadamia nuts.
18. Participant who has a condition or is in a situation that, in the investigator's opinion, may put the patient at significant risk, or may significantly interfere with the patient's participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gallo, MD, PhD, Principal Investigator — UCSD School of Medicine
Locations (1):
- University of California San Diego Dermatology Clinic, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nakatsuji T, Gallo RL, Shafiq F, Tong Y, Chun K, Butcher AM, Cheng JY, Hata TR. Use of Autologous Bacteriotherapy to Treat Staphylococcus aureus in Patients With Atopic Dermatitis: A Randomized Double-blind Clinical Trial. JAMA Dermatol. 2021 Jun 16;157(8):978-82. doi: 10.1001/jamadermatol.2021.1311. Online ahead of print. PMID 34132739

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Treatment: Autologous Microbial Transplant: Twice-daily application of Active comparators to the right and left ventral arms of patients
- Placebo Treatment: Autologous Microbial Transplant: Twice-daily application of Placebo comparators to the right and left ventral arms of patients
Period: Overall Study
Arm/Group | Active Treatment | Placebo Treatment
Started | 8 | 7
Completed | 8 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 7 | 4 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.63 (14.30) | 25.5 (12.24) | 27.85 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Relative Abundance of Staphylococcus Aureus Compared to Baseline
Description: Relative abundance of S. aureus 24 hours after initial treatment application (baseline).
Time Frame: 24 Hours
Measure: Mean (Full Range); unit: Relative abundance of S. aureus
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 8 | 6
Relative abundance of S. aureus | 0.106 [0 to 0.4] | 12.9 [1.5 to 25]

ADVERSE EVENTS:
Time Frame: 1 Month(Screening-Last Phone Call)
Arm/Group | Active Treatment | Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 1/8 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=8) | Placebo Treatment (N=6)
Rash (General disorders) | 1 (1) | 2 (2) — Rash reported in treatment area only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT03158012/Prot_SAP_000.pdf